CLINICAL TRIAL: NCT07298304
Title: The Effect of Substituting White Rice With Sorghum Rice on Pancreatic Beta-Cell Function and Insulin Resistance in Prediabetes
Brief Title: Impact of Sorghum Rice on Beta-Cell Function and Insulin Resistance in Prediabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dr. Soetomo General Hospital (Other Government)
Collaborators: Universitas Airlangga (Other)
Responsible Party: Principal Investigator, Dr. Sony Wibisono M dr., SpPD., KEMD, Principal Investigator Sony Wibisono M dr., Sp.PD., KEMD, PhD, Dr. Soetomo General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 52/EC/KEPK/FKUA/2022
Record Dates: First submitted 2025-11-25; First posted 2025-12-23 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Prediabetic State; Glucose Intolerance; Insulin Resistance; Obesity and Overweight
Keywords: Leptin; obesity; prediabetic; sorghum
MeSH Terms: conditions — Prediabetic State; Glucose Intolerance; Insulin Resistance; Obesity; Overweight

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Arm (Sorghum Group) (Experimental): 13 participants Consumed sorghum rice as a dietary substitute for 7 consecutive days Received standard lifestyle education
  Interventions: Dietary Supplement: Sorghum Rice
- Control Arm (White Rice Group): (Active Comparator): 13 participants Continued regular white rice consumption Received standard lifestyle education
  Interventions: Dietary Supplement: white rice

INTERVENTIONS:
Dietary Supplement: Sorghum Rice — Participants completely substituted all white rice intake with sorghum rice (Sorghum bicolor L.) for seven consecutive days. The amount consumed at each meal was individually calculated based on participant's daily caloric requirements. Sorghum rice was prepared using standardized cooking procedures supervised by a registered dietitian. Participants consumed sorghum rice with regular meals according to usual eating patterns. Dietary compliance was monitored daily through meal photography reviewed by research staff. Participants maintained all other usual dietary habits including portion sizes of non-grain foods, meal timing, and beverages. Both groups received identical standard lifestyle education on balanced nutrition and physical activity for prediabetes management.
  Arms: Intervention Arm (Sorghum Group)
Dietary Supplement: white rice — Participants continued habitual white rice (Oryza sativa L.) consumption for seven consecutive days without modification. The amount consumed at each meal was individually calculated based on participant's daily caloric requirements to ensure comparability with the intervention group. Participants consumed white rice with regular meals according to usual eating patterns. Dietary compliance was monitored daily through meal photography reviewed by research staff. Participants maintained all other usual dietary habits including portion sizes of non-grain foods, meal timing, and beverages. Control participants received identical standard lifestyle education on balanced nutrition and physical activity for prediabetes management.
  Arms: Control Arm (White Rice Group):

SUMMARY:
Prediabetes is a condition where blood sugar levels are higher than normal but not yet high enough to be diagnosed as diabetes. Without lifestyle changes, people with prediabetes often develop type 2 diabetes, a serious disease affecting millions worldwide. Diet plays a crucial role in preventing this progression, and replacing refined grains like white rice with whole grains may help improve metabolic health.

This study investigated whether eating sorghum rice-a nutritious whole grain rich in fiber and natural antioxidants-could affect leptin levels in people with prediabetes. Leptin is a hormone produced by fat cells that helps regulate appetite and energy use. In people with obesity and prediabetes, leptin levels are often abnormally high, which can contribute to insulin resistance and weight gain.

The investigators studied 26 police officers with prediabetes in Indonesia, randomly dividing them into two groups. One group ate sorghum rice instead of white rice for seven consecutive days, while the other group continued eating white rice. Both groups received standard education about healthy eating and exercise. The investigators measured their leptin levels before and after the week-long intervention.

Our hypothesis was that replacing white rice with sorghum rice would significantly lower leptin levels.

DETAILED DESCRIPTION:
This open-label randomized pre-post experimental study was designed to evaluate the metabolic effects of short-term sorghum rice consumption on serum leptin levels in prediabetic individuals. The study was conducted over a two-month period (March to April 2022) at the Bojonegoro Police Polyclinic and Bojonegoro Bhayangkara Hospital in East Java, Indonesia.

Rationale and Background The study addresses a critical gap in understanding dietary interventions for prediabetes management in Indonesia, where white rice consumption is a dominant dietary pattern associated with increased type 2 diabetes risk. Sorghum (Sorghum bicolor L.) represents a promising functional whole grain alternative, containing high levels of dietary fiber, resistant starch, and phenolic compounds with antioxidant properties. These bioactive components may influence adipokine profiles, particularly leptin, an adipocyte-derived hormone that plays a central role in energy homeostasis and is frequently dysregulated in prediabetic states. The study specifically targeted police officers, a population with unique physical activity patterns and occupational stress factors that may influence metabolic responses.

Twenty-six prediabetic participants were recruited through simple random sampling and randomly assigned in a 1:1 ratio to either the intervention (sorghum rice) group or the control (white rice) group, with 13 participants in each arm. The sample size was calculated using a standard formula for comparing numerical data between two independent groups, accounting for expected differences in leptin levels based on preliminary data and published literature. Randomization was performed to minimize selection bias and ensure comparable baseline characteristics between groups.

Participants in the intervention group completely substituted their regular white rice intake with sorghum rice for seven consecutive days. The sorghum rice was prepared according to standardized cooking procedures supervised by a registered dietitian to ensure consistency in preparation methods and palatability. The daily amount of sorghum or white rice consumed was individually calculated based on each participant's total daily energy requirements, determined using standard anthropometric measurements and physical activity assessments. This personalized approach ensured that participants maintained their usual caloric intake while only varying the grain type consumed.

The control group continued their habitual white rice consumption throughout the study period. Both groups received identical standardized lifestyle education sessions focusing on balanced nutrition principles and the importance of regular physical activity in prediabetes management, ensuring that any observed differences could be attributed to the grain substitution rather than differential educational interventions.

To ensure adherence to the assigned dietary intervention, participants were required to photograph each meal containing the assigned grain type and submit these images daily via mobile messaging applications. A dedicated research dietitian reviewed all submitted photographs within 24 hours to verify compliance and provide immediate feedback or guidance when needed. Participants were instructed to maintain all other aspects of their usual dietary habits, including portion sizes of non-grain foods, meal timing, and beverage consumption. This monitoring system allowed for real-time assessment of intervention fidelity while minimizing participant burden.

Anthropometric Assessments Height was measured to the nearest 0.1 centimeter using a calibrated wall-mounted stadiometer with participants standing barefoot in an erect position. Body weight was measured to the nearest 0.1 kilogram using a calibrated digital scale with participants wearing light clothing and no shoes. Body Mass Index (BMI) was calculated using the standard formula: weight in kilograms divided by height in meters squared (kg/m²). All anthropometric measurements were performed by trained research staff using standardized techniques at both baseline and follow-up assessments to ensure measurement consistency.

Biochemical Analysis Venous blood samples were collected from all participants after an overnight fast (minimum 8 hours) at baseline (day 0) and immediately following the completion of the seven-day intervention (day 7). Samples were collected in the morning (between 7:00-9:00 AM) to minimize circadian variation in hormone levels. Blood samples were allowed to clot at room temperature for 30 minutes, then centrifuged at 3,000 rpm for 10 minutes. Serum was separated and stored at -80°C until batch analysis to reduce inter-assay variability.

Serum leptin concentrations were quantified using a commercially available enzyme-linked immunosorbent assay (ELISA) kit (CAN-L-4260, Diagnostic Biochem Canada Inc., Canada) following the manufacturer's protocol. All samples were analyzed in duplicate, and the mean value was used for statistical analysis. The assay has a sensitivity of 0.5 ng/mL and demonstrates minimal cross-reactivity with other adipokines. Quality control samples were included in each assay run to ensure accuracy and precision. The change in leptin levels (delta leptin or Δ leptin) was calculated by subtracting the pre-intervention value from the post-intervention value for each participant.

Data analysis followed a pre-specified statistical plan. Continuous variables were assessed for normality using the Shapiro-Wilk test before selecting appropriate parametric or non-parametric tests. Between-group comparisons at baseline were performed to ensure group comparability. Within-group changes from baseline to post-intervention were analyzed using paired tests, while between-group differences in change scores were evaluated using independent samples tests. Subgroup analyses were conducted to explore potential effect modification by obesity status (BMI <30 vs ≥30 kg/m²). Correlation analyses examined the relationship between age and leptin change within each treatment group to identify potential demographic factors influencing treatment response. All statistical tests were two-tailed with a significance level set at α=0.05.

All study procedures were conducted in accordance with the ethical principles outlined in the Declaration of Helsinki and Good Clinical Practice guidelines. The study protocol received approval from the Health Research Ethics Committee of Health Research Ethics Committee Universitas Airlangga School of Medicine, Surabaya, Indonesia (approval number 52/EC/KEPK/FKUA/2022) prior to participant enrollment. All participants provided written informed consent after receiving detailed oral and written explanations of the study procedures, potential risks, and benefits. Participants were free to withdraw from the study at any time without penalty. Adverse events related to the dietary intervention were monitored throughout the study period through participant self-report and direct inquiry during follow-up visits.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 to 58 years
* Diagnosed with prediabetes which met one of the criteria per PERKENI 2021 as follow:
* Fasting plasma glucose 100-125 mg/dL
* 2-hour postprandial glucose 140-199 mg/dL
* HbA1c 5.7-6.4%
* Willing to comply with dietary monitoring and lifestyle instructions
* Active duty police officers

Exclusion Criteria:

* Pregnancy
* History of malignancy
* Diagnosed diabetes mellitus
* Acute infection
* Severe hepatic or renal impairment
* Current use of medication such as: glucose-lowering, corticosteroid, or anti-obesity medications

Ages: 18 Years to 58 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 26 (Actual)
Dates: Start 2022-03-01 (Actual); Primary Completion 2022-04-01 (Actual); Study Completion 2023-03-01 (Actual)

PRIMARY OUTCOMES:
Change in Serum Leptin | From Baseline to day 7
  Change in serum leptin concentration from baseline to day 7, measured using enzyme-linked immunosorbent assay (ELISA). Delta leptin (Δ leptin) calculated as the difference between post-intervention and pre-intervention leptin levels.
  Time Frame: Baseline (Day 0) and Day 7 (after 7-day intervention)Unit of Measure: Nanograms per milliliter (ng/mL)

SECONDARY OUTCOMES:
Serum Leptin Levels at Baseline | day 0, before intervention
  Baseline serum leptin concentration measured using enzyme-linked immunosorbent assay (ELISA) to establish pre-intervention values and assess differences between groupsTime Frame: Baseline (Day 0)Unit of Measure: Nanograms per milliliter (ng/mL)

CONTACTS AND LOCATIONS:
Overall Officials: Sony Wibisono Mudjanarko, dr., Sp.PD, K-EMD, PhD, Principal Investigator — Dr. Soetomo General Hospital
Locations (1):
- Soetomo General Hospital, Surabaya, East Java, Indonesia

IPD SHARING:
Plan to Share IPD: No